CLINICAL TRIAL: NCT01299779
Title: The Incidence of Hyponatremia With Two Commonly Prescribed Purgatives for Colonoscopy-Polyethylene Glycol 3350 With a Sports Drink (PEG-SD) Compared to Polyethylene Glycol 3350 With Electrolyte Solution (PEG-ELS)
Brief Title: Incidence of Hyponatremia in PEG-SD Compared to PEG-ELS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: #10C.29
Record Dates: First submitted 2010-07-12; First posted 2011-02-18 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Hyponatremia
Keywords: hyponatremia; PEG-SD; PEG-ELS
MeSH Terms: conditions — Hyponatremia | interventions — polyethylene glycol 3350; MoviPrep

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEG-ELS (Active Comparator)
  Interventions: Drug: PEG-ELS
- PEG-SD (Active Comparator)
  Interventions: Drug: PEG-SD

INTERVENTIONS:
Drug: PEG-SD — PEG-SD
  * Bisacodyl: two 5-mg tablets at 3 pm day prior
  * 1L sports drink* (labeled #1) with PEG-3350 119 gram bottle (labeled #1) at 6 pm night prior
  * 1L SD* (labeled #2) with PEG-3350 119 gram bottle (labeled #2) starting 4 hrs prior to colonoscopy
    * Same flavor, non-red Gatorade® for all patients.
  Other Names: Miralax
  Arms: PEG-SD
Drug: PEG-ELS — * 1L + 500 cc clear liquids at 6 pm night prior
  * 1L + 500 cc clear liquids starting 4 hours prior to colonoscopy
  Other Names: MoviPrep
  Arms: PEG-ELS

SUMMARY:
Objective: To compare the incidence of peri-colonoscopy hyponatremia associated with PEG 3350 + sports drink (PEG-SD) versus PEG 3350-electrolyte solution + sodium sulfate + sodium ascorbate and ascorbic acid (PEG-ELS).

Hypothesis: As compared to PEG-SD, hyponatremia occurs significantly less often with PEG-ELS.

DETAILED DESCRIPTION:
Looking at the Incidence of Hyponatremia With Two Commonly Prescribed Purgatives for Colonoscopy-Polyethylene Glycol 3350 With a Sports Drink (PEG-SD) Compared to Polyethylene Glycol 3350 With Electrolyte Solution (PEG-ELS)

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 years or older scheduled for elective outpatient colonoscopy: 8am - noon.

Exclusion Criteria:

* Unable or unwilling to consent
* Pregnant
* Breast feeding
* Significant psychiatric illness

  -> 50% colon resection
* Bowel obstruction
* History of hyponatremia (Serum sodium <135 mmol/L)
* End stage renal disease on dialysis
* History of chronic kidney disease (other than kidney stones)
* Decompensated cirrhosis, including:

  * History of bleeding due to portal hypertension (varices, gastropathy, etc) within 3 months
* Hepatic encephalopathy (not controlled with medications) within 3 months
* Clinical presence of ascites
* Active cardiac disease
* Recent myocardial infarction (<4weeks)
* Unstable angina
* Congestive heart failure NYHA Functional Class Stage III or IV
* Stage III: Marked limitation of activity. Less than ordinary activity (e.g. walking short distances, 20-100 m) causes fatigue, palpitations, dyspnea. Comfortable at rest.
* Stage IV: Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.

Exclusion Criteria (post-enrollment), from baseline labs:

* Serum creatinine > 1.5 mg/dL
* Serum potassium < 3.3 or > 5.5 mmol/L
* Serum sodium < 135 mmol/L or >150 mmol/L
* Serum calcium < 8.0 or > 11.0 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2010-06; Primary Completion 2012-05 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Development of hyponatremia in the peri-colonoscopy period | blood drawn 30 minutes post colonoscopy

SECONDARY OUTCOMES:
Development of serum electrolytes levels outside the normal range for | blood drawn 30 minutes post colonoscopy
  Sodium, chloride, potassium, calcium
Change from baseline for serum electrolytes | blood drawn 30 minutes post colonoscopy
  Sodium, chloride, potassium, calcium
Change in renal function from baseline | blood drawn pre colonoscopy and 30 minutes post colonoscopy
  Creatinine, calculated GFR
Changes in the following from baseline a. Serum vasopressin b. Serum osmolality c. Urine electrolytes and osmolality | blood drawn pre colonoscopy and 30 minutes post colonoscopy
Serum cortisol and TSH levels for only patients who develop hyponatremia | blood drawn 30 minutes post colonoscopy
Hemodynamic/volume changes at baseline and immediately prior to colonoscopy | hemodynamic measurments taken pre and post colonoscopy
  * Weight
  * Blood pressure supine and upright - systolic, diastolic
  * Pulse supine and upright
  * Development of orthostatic change: yes/no
  * Development of orthostatic symptoms - light-headed, dizzy, diaphoretic, etc.: yes/no
Adverse Events - Incidence and severity using 10-point Likert scale | 1 hour post colonoscopy assessment
  * GI - nausea, vomiting, abdominal pain, bloating
  * Light headedness
Prep Completion: <90% vs. > 90% | one time assessment pre colonoscopy
Indication for colonoscopy: Screen/Surveillance vs. Symptom | one time assessment pre colonoscopy
Assessment of independent risk factors for hyponatremia | one time assessment pre colonoscopy
  * Age
  * Sex
  * Race
  * Medications
  * Medical history
  * BMI
  * Anxiety - Beck scale
  * Fluid intake for 24 hours prior to colonoscopy (not including the prep or fluids required to accompany the prep); patients will be shown a liter container to assist with their estimate.
    i. Less than 3 Liters ii. 3-5 liters iii. More than 5 liters
Efficacy | endoscopist will evaluate during colonoscopy
  * Whole colon prep: adequate (excellent/good) vs. inadequate (fair/poor)
  * Cecal or small bowel intubation - Yes/No

CONTACTS AND LOCATIONS:
Overall Officials: David Kastenberg, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Matro R, Daskalakis C, Negoianu D, Katz L, Henry C, Share M, Kastenberg D. Randomised clinical trial: Polyethylene glycol 3350 with sports drink vs. polyethylene glycol with electrolyte solution as purgatives for colonoscopy--the incidence of hyponatraemia. Aliment Pharmacol Ther. 2014 Sep;40(6):610-9. doi: 10.1111/apt.12884. Epub 2014 Jul 28. PMID 25066025